CLINICAL TRIAL: NCT05250843
Title: TACE/HAIC Combined With Lenvatinib and Sintilimab in Neoadjuvant Therapy for Patients With Potentially High Recurrence Risk After Liver Cancer Resection: a Prospective, Randomized, Controlled Clinical Study
Brief Title: TACE/HAIC Combined With Lenvatinib and Sintilimab in Neoadjuvant Therapy for Intermediate-stage HCC
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Zhang Yingcai, doctorate, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LHuanxian
Record Dates: First submitted 2022-02-15; First posted 2022-02-22 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: Lenvatinib; TACE; PD-1
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib; sintilimab; Hepatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TACE/HAIC and Lenvatinib and PD-1(Sintilimab) before liver resection (Experimental): For patients staged BCLC B/C,TACE/HAIC combined with Lenvatinib and Sintilimab will be conducted as neoadiuvent therapy before liver resection
  Interventions: Procedure: TACE/HAIC; Drug: Lenvatinib; Drug: Sintilimab
- Direct surgery group (Active Comparator): After being diagnosed with hepatocellular carcinoma, surgery will be immediately performed.
  Interventions: Procedure: liver resection

INTERVENTIONS:
Procedure: TACE/HAIC — Within 1-3 days of lenvatinib and sintilimab, start Transarterial chemobolization treatment or FOLFOX-based chemotherapy infusion,after three months,patients who achieved partial response (PR) or minor response (MR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and were assessed as eligible for R0 resection go on to undergo surgical resection.
  Arms: TACE/HAIC and Lenvatinib and PD-1(Sintilimab) before liver resection
Drug: Lenvatinib — Participants received lenvatinib capsules 8mg for patients weight <60kg, or 12mg for patients weight more than 60Kg.
  Arms: TACE/HAIC and Lenvatinib and PD-1(Sintilimab) before liver resection
Drug: Sintilimab — Sintilimab Injection will be administered every three weeks (200mg) until surgery or disease progression.
  Arms: TACE/HAIC and Lenvatinib and PD-1(Sintilimab) before liver resection
Procedure: liver resection — liver resection is feasible after evaluation by the liver cancer surgery expert group
  Arms: Direct surgery group

SUMMARY:
The purpose of the study is to observe the effect of TACE/HAIC combined with lenvatinib and sintilimab as a neoadjuvant therapy before liver resection in preventing the recurrence in high-risk patients with hepatocellular carcinoma.

DETAILED DESCRIPTION:
For patients with hepatocellular carcinoma staged BCLC B/C(intermediate hepatocellular carcinoma)，TACE is a widely used treatments .However ,The efficacy of TACE in intermediate hepatocellular carcinoma is not very satisfactory.A series of study demonstrated that direct hepatectomy has better prognosis compared with TACE for these intermediate hepatocellular carcinoma patients.Despite of this ,The high recurrence risk, high probability of surgical complications, and poor treatment effect after recurrence of intermediate hepatocellular carcinoma after direct surgical treatment is a still a tough problem to be solved.Recently, investigators have showed that hepatic arterial infusion of FOLFOX-based chemotherapy (HAIC) was safe and efficient for advanced HCC patients. The combination of TACE with HAIC (TACE-HAIC) was proved to increase the local doses of chemotherapeutic agents in the liver .In addition, Lenvatinib was proved non-inferior to sorafenib in overall survival in advanced hepatocellular carcinoma, and Programmed Cell Death Protein-1 (PD-1) antibody was effective and tolerable in patients with advanced hepatocellular carcinoma.In this context，for those patients with potentially high recurrence risk after liver resection, the investigators carried out this prospective randomized control to demonstrate the superiority of TACE/HAIC combined with PD-1 antibody and lenvatinib as a neoadjuvant therapy before liver resection over direct hepatectomy.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age 18-70 years old, gender is not limited.
* 2)The diagnosis of HCC was based on the diagnostic criteria for HCC used by the European Association for the Study of the Liver (EASL).
* 3)Patients must have at least one tumor lesion that can be accurately measured.
* 4)Conform to any of the following criteria (1) multiple nodules >3; (2) ≥2 nodules, any of which is >3 cm; (3) invasion of the portal vein or hepatic vein.
* 5)According to the 2022 edition of the Chinese guidelines for the diagnosis and treatment of primary liver cancer, one-stage liver cancer resection is feasible after evaluation by the liver cancer surgery expert group
* 6)No previous anti-HCC treatment.
* 7)Eastern Co-operative Group performance status 2 or less.
* 8)Liver function: Child's A or B (score < 7).

Exclusion Criteria:

* 1)Patients with definite tumor thrombus and distant metastasis in the main portal vein and inferior vena cava;
* 2) Allergy to the components of intervention-related drugs such as lipiodol and chemotherapeutic drugs;
* 3) Local treatment (including intervention, surgery, ablation, etc.) and systemic treatment (chemotherapy, targeted drugs and immune checkpoint inhibitors, etc.) for liver cancer within the past 2 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free Survival | 12 months
  Time from the start of liver resection until tumor recurrence or death (from any cause).

SECONDARY OUTCOMES:
Adverse effects | 12 months
  Frequency and severity of adverse effects as defined by CTCAE version 5

CONTACTS AND LOCATIONS:
Locations (1):
- Third Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No